CLINICAL TRIAL: NCT04575727
Title: Exploratory Evaluation of [11C]MPC6827 Pharmacokinetics With Positron Emission Tomography (PET)
Brief Title: Exploratory Evaluation of [11C]MPC6827
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Columbia University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: AAAS4926
Record Dates: First submitted 2020-09-29; First posted 2020-10-05 (Actual); Last update posted 2025-04-13 (Actual); Status verified 2025-04

CONDITIONS: Neurodegenerative Diseases; Alzheimer Disease; Amyotrophic Lateral Sclerosis
Keywords: [11C]MPC6827
MeSH Terms: conditions — Neurodegenerative Diseases; Alzheimer Disease; Amyotrophic Lateral Sclerosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Health Volunteers (Experimental): In the first stage, five healthy human subjects will receive a microdose (10 µg) of [11C]MPC6827, immediately followed by whole body PET/CT to determine dosimetry and perform an initial safety evaluation of the radiotracer. A dose of 20 mCi [11C]MPC6827 will be administered and serial whole body PET scans will be acquired up to 2 hours post injection.
  Interventions: Drug: [11C]MPC6827
- Patients with Neurodegenerative Disorders (Experimental): Up to 30 patients with neurodegenerative disorders will receive a microdose (10 µg) of [11C]MPC6827 and be imaged dynamically for up to 90 minutes using PET/CT for research purposes.
  Interventions: Drug: [11C]MPC6827

INTERVENTIONS:
Drug: [11C]MPC6827 — Subjects will receive a microdose ( 10 µg) of [11C]MPC6827 (dose of 20 mCi)
  Other Names: [11C]MPC

SUMMARY:
This is a phase 0 study that will enable an assessment of biodistribution and estimation of absorbed dose in humans based on data collected from five healthy volunteers, which is typically the minimum number required by the FDA for first-in-human studies to assess dosimetry of a new tracer. The evaluation of the brain imaging of thirty additional subjects in the 2nd part of the study will lead to a descriptive assessment of the targeting and pharmacokinetics of MPC6827 in the brain and between normal and diseased brain.

DETAILED DESCRIPTION:
Neurodegenerative diseases are conditions where the brain cells break down, causing mental and/or physical impairment. Alzheimer's Disease is a neurodegenerative disorder that affects millions of individuals and causes irreversible memory loss and cognitive impairment. Amyotrophic lateral sclerosis is also and incurable disorder that causes patients irreversible paralysis, which results in death due to inability to breath and suffocation. These disease have been shown to be associated with abnormalities in an important scaffolding called microtubules, a cellular structure that help support the shape of the cells. This study will explore an experimental imaging test to see if it can be used to help doctors identify early microtubule changes. The test involves the injection of a radioactive compound that has been shown to go to cells and bind to microtubules. Special cameras called Positron Emission Tomography (PET)/CT cameras will be used to allow doctors to view where the radioactive compound goes in the body, as this is the first time this radiolabeled agent is being used in humans. In this study, doctors will give the new compound to up to five healthy volunteers to see where it goes in the body of people who presumable have normal microtubule function. Then doctors will give [11C]MPC6827 to up to 30 additional subjects (healthy controls and patients with Alzheimers Disease or ALS) to focus on imaging the brain for extended times. The research-imaging drug in this study is [11C]MPC6827. The radioactive drug in this study is experimental, meaning it is not approved by the FDA and can only be used in research studies.

ELIGIBILITY:
Inclusion Criteria (Healthy Volunteers)

1. All volunteers must be 18 years of age or older, able to read, understand and voluntarily sign and informed consent document.
2. Volunteers must have no current medical history of brain disease
3. Negative pregnancy test if female of childbearing potential.
4. Women of childbearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry for the duration of study participation.

Inclusion Criteria (Alzheimer's Disease or ALS)

1. All volunteers must be 18 years of age or older, able to read, understand and voluntarily sign and informed consent document.
2. Subjects must have a diagnosis of Alzheimer's Disease or ALS for which they are under a physician's care.
3. Subjects must have a negative pregnancy test if female of childbearing potential
4. Women of childbearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry for the duration of the study participation.

Exclusion Criteria:

1. Participants with evidence of brain disease other than ALS or Alzheimer's Disease at the time of enrolment up to agent administration are to be excluded from the study.
2. Concomitant medication use that, in the judgement of the investigator, would make the participant inappropriate for enrolment.
3. Severe concurrent disease, infection, or medical co-morbidity that, in the judgement of the investigator, would make the participant inappropriate for enrolment.
4. Participants who are receiving other investigational radiation drugs.
5. Women who are pregnant or breast feeding.
6. Subjects who are unable to tolerate PET/CT imaging

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2021-01-08 (Actual); Primary Completion 2024-06-21 (Actual); Study Completion 2024-06-21 (Actual)

PRIMARY OUTCOMES:
Biodistribution of [11C]MPC6827 | up to 48 hours from injection
  Total body residence time and visual examination of whole body PET/CT images will be used to determine biodistribution of [11C]MPC6827.
Estimation of clearance of [11C]MPC6827 | Up to 48 hours from injection
  Serial venous blood draws (about 5 ml per sample) will be taken for estimation of clearance of [11C]MPC6827.

CONTACTS AND LOCATIONS:
Overall Officials: Akiva Mintz, MD, Principal Investigator — Columbia University
Locations (1):
- Cuimc / Nyp, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No
Final data analysis and conclusion will be submitted to scientific journals and made available for publication.